CLINICAL TRIAL: NCT04892537
Title: Coronary Sinus Reducer Objective Impact on Symptoms, MRI Ischaemia and Microvascular Resistance
Acronym: ORBITA-COSMIC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Imperial College London (Other)
Collaborators: Medical Research Council (Other Government); Imperial College Healthcare Nissen Fund (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20HH6457; MR/V001620/1 (Other Grant/Funding Number: Medical Research Council)
Record Dates: First submitted 2021-04-30; First posted 2021-05-19 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2023-10

CONDITIONS: Refractory Angina
MeSH Terms: conditions — Angina Pectoris

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CSR (Active Comparator): Coronary Sinus Reducer implantation
  Interventions: Device: Coronary Sinus Reducer
- Placebo (Placebo Comparator): Placebo procedure
  Interventions: Procedure: Placebo Procedure

INTERVENTIONS:
Device: Coronary Sinus Reducer — Coronary Sinus Reducer implantation according to standard clinical protocols
  Other Names: CSR
  Arms: CSR
Procedure: Placebo Procedure — A placebo procedure involving venous sheath implantation in the right internal jugular vein without proceeding to CSR implantation
  Arms: Placebo

SUMMARY:
ORBITA-COSMIC is a randomised, double-blinded, placebo controlled trial of the coronary sinus reducer (CSR). The investigators will compare the effects of CSR versus placebo on myocardial perfusion on MRI, exercise time and symptoms in 50 participants with refractory angina and ischaemia.

ELIGIBILITY:
Inclusion Criteria:

* Stable coronary artery disease (CAD) not eligible for percutaneous coronary intervention (PCI) or coronary artery bypass graft surgery (CABG)
* Evidence of ischaemia on stress perfusion CMR
* Angina - Canadian Cardiovascular Society Class II-VI on maximal medical therapy

Exclusion Criteria:

* Age<18 years
* Pregnancy
* Inability to consent
* Recent acute coronary syndrome (3 months)
* Recent revascularisation (6 months)
* Permanent pacemaker or defibrillator leads in the right heart
* Severe left ventricular impairment (<25%)
* Indication for cardiac resynchronisation therapy (CRT)
* Right atrial pressure ≥15mmHg
* Life expectancy <1 year
* Severe renal impairment (eGFR<15)
* Contraindication to CMR
* Contraindication to adenosine
* Ischaemia isolated to inferior wall
* Ongoing participation in a separate interventional study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-05-21 (Actual); Primary Completion 2024-01 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Myocardial Blood Flow | 6 months
  On cardiac MRI, with adenosine stress, millilitres/gram/minute

SECONDARY OUTCOMES:
Myocardial perfusion reserve (MPR) in ischaemic segments, non ischaemic segments and global MPR | 6 months
  On cardiac MRI
Rest myocardial blood flow (MBF) in ischaemic segments, non ischaemic segments and global rest MBF | 6 months
  On cardiac MRI, millilitres/gram/minute
Stress myocardial blood flow (MBF) in ischaemic segments, non ischaemic segments and global stress MBF | 6 months
  On cardiac MRI, millilitres/gram/minute
MPR in ischaemic segments with inferior and inferoseptal segments excluded | 6 months
  On cardiac MRI
MBF in ischaemic segments with inferior and inferoseptal segments excluded | 6 months
  On cardiac MRI, millilitres/gram/minute
Endocardial:epicardial ratio of stress MBF | 6 months
  On cardiac MRI
Endocardial:epicardial ratio of rest MBF | 6 months
  On cardiac MRI
Endocardial:epicardial ratio of MPR | 6 months
  On cardiac MRI
Myocardial strain | 6 months
  On cardiac MRI
Myocardial scar burden | 6 months
  On cardiac MRI
Episodes of angina component of angina symptom score | 6 months
  Daily episodes recorded on ORBITA-COSMIC smartphone application
Canadian Cardiovascular Society Class | 6 months
  On a scale from 0-4 with higher scores indicating more severe angina
Angina symptom score | 6 months
  Derived from ORBITA-COSMIC smartphone application
Seattle Angina Questionnaire (SAQ) Angina Frequency | 6 months
  On a scale from 0-100, with higher scores indicating better outcomes
SAQ Angina Physical Limitation | 6 months
  On a scale from 0-100, with higher scores indicating better outcomes
SAQ Quality of Life | 6 months
  On a scale from 0-100, with higher scores indicating better outcomes
SAQ Treatment Satisfaction | 6 months
  On a scale from 0-100, with higher scores indicating better outcomes
SAQ Angina Stability | 6 months
  On a scale from 0-100, with higher scores indicating better outcomes
Euro-Qol (EQ-5D-5L) descriptive system | 6 months
  Index derived from 5 question domains, with higher scores indicating better quality of life
Euro-Qol (EQ-5D-5L) visual analogue scale | 6 months
  Visual analogue scale from 0-100 with 100 indicating better quality of life
Angina related quality of life rated by the MacNew questionnaire | 6 months
  On a scale from 1-7 with higher scores indicating better quality of life
Treadmill Exercise Time | 6 months
  Modified Bruce Protocol
Absolute coronary flow on pressure/temperature wire assessment | 6 months
  millilitres per minute
Absolute coronary resistance on pressure/temperature wire assessment | 6 months
  mmHg/(L/min)
Microvascular resistance reserve on pressure/temperature wire assessment | 6 months
Coronary flow reserve (CFR) on pressure/temperature wire assessment | 6 months
Index of microcirculatory resistance on pressure/temperature wire assessment | 6 months
CFR assessed by a pressure and doppler sensor wire | 6 months

CONTACTS AND LOCATIONS:
Locations (5):
- United Kingdom (5):
  - Basildon and Thurrock Hospitals NHS Foundation Trust, Basildon
  - Royal Bournemouth Hospital, Bournemouth
  - Imperial College Healthcare NHS Trust, London
  - St George's Hospital, London
  - The Royal Brompton Hospital, London

REFERENCES:
- [Derived] Foley MJ, Rajkumar CA, Ahmed-Jushuf F, Simader FA, Chotai S, Pathimagaraj RH, Mohsin M, Salih A, Wang D, Dixit P, Davies JR, Keeble TR, Cosgrove C, Spratt JC, O'Kane PD, De Silva R, Hill JM, Nijjer SS, Sen S, Petraco R, Mikhail GW, Khamis R, Kotecha T, Harrell FE, Kellman P, Francis DP, Howard JP, Cole GD, Shun-Shin MJ, Al-Lamee RK. Coronary sinus reducer for the treatment of refractory angina (ORBITA-COSMIC): a randomised, placebo-controlled trial. Lancet. 2024 Apr 20;403(10436):1543-1553. doi: 10.1016/S0140-6736(24)00256-3. Epub 2024 Apr 8. PMID 38604209
- [Derived] Foley MJ, Rajkumar CA, Ahmed-Jushuf F, Simader F, Pathimagaraj RH, Nijjer S, Sen S, Petraco R, Clesham G, Johnson T, Harrell FE Jr, Kellman P, Francis D, Shun-Shin M, Howard J, Cole GD, Al-Lamee R. A double-blind, randomised, placebo-controlled trial of the coronary sinus Reducer in refractory angina: design and rationale of the ORBITA-COSMIC trial. EuroIntervention. 2024 Feb 5;20(3):e216-e223. doi: 10.4244/EIJ-D-23-00567. PMID 38214677